CLINICAL TRIAL: NCT01947231
Title: Randomized Controlled Trial of Global Postural Re-education vs. Standard Manual Physical Therapy for Non-specific Chronic Neck Pain With Cross-over
Brief Title: GPR vs Manual PT for Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, paolo pillastrini, Associate Professor and President of Baccaluareate Course in Physiotherapy, University of Bologna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2436/2013
Record Dates: First submitted 2013-09-03; First posted 2013-09-20 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Nonspecific Chronic Neck Pain
Keywords: neck pain; chronic; Global Postural Re-education; manual therapy; physical therapy
MeSH Terms: conditions — Neck Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Global Postural Re-education (Experimental): Global Postural Re-education is delivered in a single treatment session each week for nine weeks.
  Interventions: Other: Global Postural Re-education
- Standard manual physical therapy (Active Comparator): Standard manual physical therapy is delivered in a single treatment session each week for 9 weeks.
  Interventions: Other: Standard manual physical therapy

INTERVENTIONS:
Other: Global Postural Re-education — Global Postural Re-education is a physical therapy method comprising a series of gentle active movements, implemented by the therapist using manual contacts and verbal commands, to promote postural symmetry.
  Arms: Global Postural Re-education
Other: Standard manual physical therapy — Standard manual physical therapy in this study involves a combination of exercises, pompage (gentle manual techniques of distraction and articulation of a joint), anterior-posterior mobilizations as described by Maitland, and massage that have been selected to meet the needs of each individual patient.
  Arms: Standard manual physical therapy

SUMMARY:
Effective treatment for nonspecific chronic neck pain is a clinical challenge. Patients will be randomized into two groups to compare the outcomes of Global Postural Re-education (GPR) with standard manual physical therapy on with respect to pain, function, kinesiophobia, range of motion, perceived effect, and satisfaction.

DETAILED DESCRIPTION:
These study will use two groups: one to receive GPR which is a systematic method of addressing musculoskeletal pain and related functional deficits and the other to receive "usual care" manual PT which will be individualized to the patient's condition. Usual care will include techniques commonly used in clinical practice selected by the physical therapist after initial examination. After nine weeks of treatment, baseline measures will be re-evaluated. After conclusion of the first phase of the study, patients who were randomized to the "usual care" group will cross-over and receive GPR.

ELIGIBILITY:
Inclusion Criteria:

-nonspecific neck pain lasting at least 3 months

Exclusion Criteria:

* acute or subacute cervical pain
* specific or known cause of pain
* central or peripheral neurological signs
* systemic pathology
* rheumatologic pathology
* neuromuscular pathology
* cognitive impairment
* surgical intervention in the last 6 months prior to study
* physical therapy treatment in the last 6 months prior to study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Pain | 9 weeks after start of intervention
  The investigators assessed this outcome with a Visual Analogue Scale (VAS).
Cervical Functional Limitations | 9 weeks after start of intervention
  The investigators assessed this outcome with the Neck Disability Index.

SECONDARY OUTCOMES:
Kinesiophobia | 9 weeks after start of intervention
  The investigators assessed this outcome with the Tampa Scale of Kinesiophobia.
Cervical Range of Motion | 9 weeks after start of intervention
  The investigators assessed this outcome with the CROM-Deluxe which is an inclinometer that is placed on the subject's head to measure cervical range of motion.
Self-reported Global Effect of the Intervention | 9 weeks after start of intervention
  The investigators assessed this outcome with a Global Perceived Effect scale which measures the subject's self-reported improvement or deterioration following the intervention.
Patient Satisfaction | 9 weeks after start of intervention
  The investigators assessed this outcome with the Physical Therapy Patient Satisfaction Questionnaire - Italian Version which has established psychometric properties.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pillastrini, Principal Investigator — University of Bologna
Locations (1):
- Policlinico S. Orsola-Malpighi, Bologna, Emiglia-Romagna, Italy